CLINICAL TRIAL: NCT05951361
Title: Evaluation of Diode Laser and Topical Steroid Therapy in the Treatment of Erosive Oral Lichen Planus (A Randomized Controlled Clinical Trial)
Brief Title: Evaluation of Diode Laser and Topical Steroid Therapy in the Treatment of Erosive Oral Lichen Planus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0369-01/2022
Record Dates: First submitted 2023-06-28; First posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-06

CONDITIONS: Erosive Oral Lichen Planus
MeSH Terms: interventions — Lasers, Semiconductor

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: the patients were randomly assigned to avoid bios.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kenacourt-A Orabase (Active Comparator): the patients in this group received steroid therapy" Kenacourt-A Orabase" three times daily for 4 weeks.
  antifungal drug "miconazole oral gel" once daily for 1 week
  Interventions: Drug: 0.1% topical triamcinolone Acetonide preparation "Kenacourt-A Orabase"
- 980nm Diode Laser (Active Comparator): the patients received 980 nm diode laser treatment 300 mW, non-contact mode up to 10 sessions
  Interventions: Device: 980nm Diode Laser

INTERVENTIONS:
Device: 980nm Diode Laser — 300 mW, 4 J/cm2, 2mm non-contact mode up to 10 sessions
  Arms: 980nm Diode Laser
Drug: 0.1% topical triamcinolone Acetonide preparation "Kenacourt-A Orabase" — three times daily for 4 weeks
  Other Names: Kenacourt-A Orabase
  Arms: Kenacourt-A Orabase

SUMMARY:
this study evaluates the effect of diode laser in treatment of oral lichen planus.

DETAILED DESCRIPTION:
44 patients with erosive oral lichen planus were included in the study and divided into 2 equal groups. Group I received topical steroid therapy three times daily for 4 weeks and antifungal oral gel once daily for 1 week. Group II received 980nm Diode Laser 300 mW, up to 10 sessions.

ELIGIBILITY:
Inclusion Criteria:

* Patient histologically diagnosed with erosive OLP based on WHO modified criteria 2003.
* Presence of painful erosive OLP lesions diagnosed by biopsy

Exclusion Criteria:

* Pregnant or breast-feeding women
* Patients currently treated for cancer with Chemotherapy or Radiotherapy
* Patient currently on Corticosteroid therapy or had this treatment on the past 3 months
* Those who had used Anti-inflammatory drugs topical or systemic in the last month
* the use of drugs related to Oral Lichenoid Lesions
* Presence of Amalgam restorations near the OLP lesions
* dysplasia in histopathological examination
* uncontrolled systemic diseases
* physical or mental abnormality which would interfere with or be affected by the study procedure
* Patients with skin lesion

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-02-10 (Actual); Study Completion 2023-04-10 (Actual)

PRIMARY OUTCOMES:
change of pain from the base line to 12 weeks follow-up | base line, 6weeks and 12 weeks
  Vas is one way to express pain into a numerical value where 0 means no pain and 10 means worst pain ever

SECONDARY OUTCOMES:
change of clinical score of the lesion from the base line to 12 weeks follow-up | base line, 6weeks and 12 weeks
  The size of the lesion is monitored where score 0 no lesions, score 1 : mild white striation only, score 2 : white striation with erythematous area < 1 cm 2, score 3 : white striation with erythematous area > 1 cm 2, score 4 : white striation < 1 cm2, score 5 : white striation with erosive area > 1 cm2.

OTHER OUTCOMES:
change in lipid peroxidation marker malondialdehyde from the base line to 12 weeks follow-up o 10 points VAS | base line, 6weeks and 12 weeks
  malondialdehyde is a strong marker for lipid peroxidation that can be measured in saliva to assess the effect of the treatment in oral lichen planus

CONTACTS AND LOCATIONS:
Overall Officials: Naguiba Mahmoud, Prof, Study Director — department of oral medicine, faculty of dentistry
Locations (1):
- Faculty of Dentistry, Department of Oral Medicine, Periodontology, Oral Diagnosis and Oral Radiology, Alexandria, Alexandria Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Access to the data may be extended beyond the initial 24-month period upon request and approval, which will also be evaluated on a case-by-case basis.
Supporting Information: Study Protocol, SAP
Time Frame: The submission of data requests can commence nine months after the article has been published, and the data will be available for up to 24 months. Extensions will be reviewed on a case-by-case basis.
Access Criteria: Qualified researchers who are conducting independent scientific research may request access to trial IPD. Upon review and approval of a research proposal and Statistical Analysis Plan (SAP), and the execution of a Data Sharing Agreement (DSA), access will be granted. For additional information or to request access, please contact the data provider. Approval for the extension of access beyond the initial 24-month period will also be considered on a case-by-case basis.

REFERENCES:
- [Background] Cafaro A, Arduino PG, Massolini G, Romagnoli E, Broccoletti R. Clinical evaluation of the efficiency of low-level laser therapy for oral lichen planus: a prospective case series. Lasers Med Sci. 2014 Jan;29(1):185-90. doi: 10.1007/s10103-013-1313-6. Epub 2013 Apr 3. PMID 23549680
- [Background] Dillenburg CS, Martins MA, Munerato MC, Marques MM, Carrard VC, Sant'Ana Filho M, Castilho RM, Martins MD. Efficacy of laser phototherapy in comparison to topical clobetasol for the treatment of oral lichen planus: a randomized controlled trial. J Biomed Opt. 2014 Jun;19(6):068002. doi: 10.1117/1.JBO.19.6.068002. PMID 24887747
- [Derived] Mohamed RK, Elsayed NM, Mahmoud SA, Gaweesh YY. Photobiomodulation versus corticosteroid in the management of erosive oral lichen planus: a randomized controlled clinical trial. BMC Oral Health. 2024 Feb 17;24(1):246. doi: 10.1186/s12903-024-03976-6. PMID 38365694

DOCUMENTS (1):
  • Study Protocol (2022-02-07): https://cdn.clinicaltrials.gov/large-docs/61/NCT05951361/Prot_000.pdf